CLINICAL TRIAL: NCT05142956
Title: Smoking Increases the Risk of Postoperative Wound Complications: a Propensity Score-matched Cohort Study
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chao-Shun Lin, Attending physician of anesthesiology, clinical professor, Taipei Medical University Hospital
Other Study IDs: soonlin0001
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Wound Complication; Smoking; Postoperative Complications
Keywords: Smoking; Postoperative wound complications
MeSH Terms: conditions — Smoking; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smokers: Current smokers are defined as cigarettes smoking within one year before surgery.

SUMMARY:
Cigarette smoking is associated with surgical complications, including wound healing and surgical site infection. However, the association between smoking status and postoperative wound complications is not completely understood. Our objective is to investigate the effect of smoking on postoperative wound complications for major surgeries.

DETAILED DESCRIPTION:
Smoking at the time of surgery is recognized as a risk factor for cardiovascular, respiratory, and wound-related perioperative complications. Wound-related complications can prolong hospital stays, increase hospital resource utilization, and pose an obvious threat to patient recovery. A brief statement on perioperative smoking cessation about smoking impacting wound healing was published by the American Society of Anesthesiologists' Task Force on Smoking Cessation. Recently, a consensus statement on perioperative smoking cessation by Society for Perioperative Assessment and Quality Improvement (SPAQI) mentioned that smoking cessation should be done as soon as practicable with surgical scheduling. More extended abstinence is associated with lower rates of wound healing complications.

Several studies have described smoking harms wound healing in specific operations, such as plastic surgery, breast surgery, gastrointestinal surgery, and hip surgery. They found surgical site infection and wound delayed healing more frequently in smokers. But in a few small studies and some surgery, conflicting results were found. Besides, risk factors associated with wound complications include infection, smoking, aging, malnutrition, immobilization, diabetes, vascular disease, and immunosuppressive therapy.

This study aims to determine the impact of smoking on wound complications for all kinds of major surgeries. To clarify the risks, our study uses the updated National Surgical Quality Improvement Program (NSQIP) database to find if patients who were active smokers are more likely to have wound-related complications postoperatively. We hypothesized that the active smoking population will have increased infectious complications and wound dehiscence compared with the nonsmoking population.

ELIGIBILITY:
Inclusion Criteria:

* From NSQIP dataset, patients with complete information for baseline parameters and without preoperative open wound infections

Exclusion Criteria:

* Incomplete information of baseline parameters, and with preoperative wound infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical cases from 2013-2018 NSQIP dataset
Sampling Method: Non-Probability Sample
Enrollment: 1150000 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
wound complications | within 30 days after the primary procedure
  surgical site infection and wound disruption

SECONDARY OUTCOMES:
pulmonary complications | within 30 days after the primary procedure
  reintubation or ventilator > 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Shun Lin, PhD, Study Chair — Department of Anesthesiology, Taipei Medical University Hospital, 252 Wuxing St., Taipei 110 Taiwan
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan